CLINICAL TRIAL: NCT03666806
Title: Preventing Stroke Triggers in Children With Sickle Cell Anaemia in Mulago Hospital, Kampala (PREST ): a Randomized Control Trial
Acronym: PREST
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Makerere University (Other)
Responsible Party: Principal Investigator, College of Health Sciences, makchs, Makerere University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: #REC REF 2018-108
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Preventing Stroke in Sickle Cell Anaemia
Keywords: Sickle cell anaemia, stroke, preventing, children, Uganda
MeSH Terms: conditions — Anemia, Sickle Cell; Stroke | interventions — Influenza Vaccines

STUDY DESIGN:
Intervention Model Description: Randomized double blinded parallel control study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participant and the study team will both be masked to which arm the participant will be assigned. Blinding will be achieved by use of a placebo that has similar characteristics as the influenza vaccine i.e. as the vaccine, the placebo will be formulated and packaged as an injectable placebo. In addition, on enrollment, the participants will be informed by the study team that their assignment to a study arm is completely random and unknown to the study team. The study nurse will pick the study drug from the pharmacist to be used for each participant after the randomization code has been revealed. The randomization code on the study drug will have to be the same as the code in the envelope. Lastly, the envelopes will be kept off site with the statistician who will deliver them every morning before the clinic opens.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Influenza vaccine (Experimental): Influenza vaccine: An inactivated influenza vaccine (split virion) shall be used during the study. The product information is attached as an appendix to the proposal. Brief description of the type of influenza vaccine to be used for the study, mechanism of action, dose justification, efficacy, safety and its use in the population.
  Interventions: Biological: Influenza vaccine
- Normal saline (Placebo Comparator): Placebo: Placebo will be normal saline which shall be prepared by the pharmacist for injection by the immunization nurse in a similar syringe as the investigational product.
  Interventions: Biological: Influenza vaccine

INTERVENTIONS:
Biological: Influenza vaccine — The randomized FLUVACS trial demonstrated the benefits of influenza vaccination in the prevention of cardiovascular death. In the VIPS study the risk for acute ischaemic stroke (AIS) in children increased by 6-fold compared to the baseline population. It was postulated that infections and in particular upper respiratory tract infections acts as a stroke trigger in a child who is otherwise predisposed to stroke and why it would occur at a particular point in that child's life. It should be noted that major infections such as meningitis have been causes of stroke while this study has shown that minir infections can also act as a trigger for stroke in adults

SUMMARY:
Sickle cell anaemia (SCA) is a common hereditary haemoglobin disorder in Africa. World wide it is estimated that about 300,000 newborns are born every year. Of which 75% of them live in Sub-saharan Africa (SSA). In Uganda, about 15,000 babies are born with sickle cell disease per year.

In Uganda, the stroke prevalence was found to be 6.2% in children admitted to the National referral hospital in Kampala. Notable between 21 to 30% of these children presented with co-morbidities such as anaemia, bacteraemia and painfull crisis. Stroke in SCA is mediated by several mechanism such as cellular adhesions, inflammatory markers, hemolysis associated oxidative stress and hemostatic activation. Stroke in SCA is primarily a large vessel stroke and the mechanisim state above lead to a narrowing of the lumen of the cerebral arteries Arterial ischaemic stroke which occurs frequently in children with SCA has been associated with bacterial infections. Recent studies have shown that minor infections such as flu like infections can play a critical role in the trigger of stroke in children.

Our hypothesis is that viral flu infections is a key trigger for the risk of stroke in children with SCA. Our objective is to prevent the occurrence of flu illnesses in children with SCA thereby reducing the risk for stroke in our population of children with SCA.

Methods: A randomized controlled double blinded study Study site: The study will be conducted at the Sickle Cell Clinic (SCC), Mulago Hospital. Inclusion criteria: will be ;age between 2 years and 12 years;All children whose parents will have consented and those above 7years will have to assent. Exclusion criteria: all children with previous strokes; children who have acute illness and are not clinically stable; any child with previous documented adverse event following immunization (AEFI).

Sample Size: Using Open EPI calculator for cohort studies we calculated a total sample size of 136 participant to achieve our objective. Using a 95% confidence interval, power of 80% and an unexposed outcome of 25% (4) using a ratio of 1:1. Each arm will have 68 participants. With anticipated 10% loss to follow up a total sample size of 150 with each arm having 75 participants.

Study utility: Globally, stroke triggers have been recently identified independent of the existing risk factors such as high cerebral velocity speeds on TCDs. Flues like illnesses have been reported to be stroke triggers in children with arterial ischaemic strokes worldwide.This study may influence the role of influenza vaccination in the prevention of stroke triggers in children with sickle cell anaemia. It will also add to the existing modalities which have helped to reduce the incidence of stroke amongst this high risk group of children with

DETAILED DESCRIPTION:
Preventing Stroke Triggers in Children with Sickle Cell Anaemia in Mulago Hospital, Kampala (PREST): A Randomized Control Trial

Principal Investigator: Deogratias Munube ( MBChB, MMed) Department of Paediatrics and Child Health

Mentor: Prof . James.K. Tumwine (MBChB, MMed, PhD) Prof . Grace Ndeezi (MBChB, MMed, PhD)

Research hypothesis: Our hypothesis is that viral flu infections is a key trigger for the risk of stroke in children with SCA. Our objective is to prevent the occurrence of flu illnesses in children with SCA thereby reducing the risk for stroke in our population of children with SCA.

Rational for research: Globally, stroke triggers have been recently identified independent of the existing risk factors such as high cerebral velocity speeds on TCDs. Flues like illnesses have been reported to be stroke triggers in children with arterial ischaemic strokes worldwide. This study may influence the role of influenza vaccination in the prevention of stroke triggers in children with sickle cell anaemia. It will also add to the existing modalities which have helped to reduce the incidence of stroke amongst this high risk group of children with

Methods: Study design: This will be a randomized controlled double blinded study Study site: The study will be conducted at the Sickle Cell Clinic (SCC), Mulago Hospital.

Study population: The study will include individuals with Sickle cell anaemia attending the sickle cell clinic services at Mulago National Referral Hospital.

Inclusion criteria: Age between 2 years and 12 years; all children whose parents will have consented and those above 7years will have to assent Exclusion criteria: All children with previous strokes; Children who have acute illness and are not clinically stable; any child with previous documented adverse event following immunization (AEFI).

Sample Size: Using Open EPI calculator for cohort studies we calculated a total sample size of 136 participants to achieve our objective. Using a 95% confidence interval, power of 80% and an unexposed outcome of 25% (4) using a ratio of 1:1. Each arm will have 68 participants. With anticipated 10% loss to follow up a total sample size of 150 with each arm having 75 participants.

The following will be done to achieve a randomized control trial:

1. Randomization
2. Blinding
3. Study variables:

Primary outcome: Incidence of stroke: The incidence of stroke is defined as the occurrence of a focal neurological deficit in a child lasting at least 24 hours if it has a vascular basis during the study period. Each child suspected to have stroke will have a brain cranial tomography (CT) scan done to confirm the diagnosis. This diagnosis will then be adjudicated by a team comprising of a pediatrician, neurologist and a radiologist.

Secondary outcomes: The levels of inflammatory markers VCAM-1 and gene profile IL4R 503P locus: blood will extracted from a participant by veni-puncture every 6 months and whenever a participant comes to the clinic when ill or is admitted, Acute chest syndrome, Pneumonia.

Trans-cranial Doppler scan speeds: a TCD will be performed for each participant every 6 months and whenever the participant is admitted or comes to the clinic when ill. The speeds will be noted.

Investigational products: influenza vaccine: An inactivated influenza vaccine (split virion) shall be used during the study. The product information is attached as an appendix to the proposal.

Study product acquisition: The product will be acquired from Laborex pharmaceutical, Sure House, Bombo road, Kampala.The vaccine is an injectable packaged in a vial Preparation, administration and dosage of the influenza vaccine to be used for the study Placebo: Placebo will be the sterile water for injection which shall be withdrawn from a vial for each participant.

Recruitment procedures: All children with SCD from 2 to 12 years presenting at the sickle cell clinic will be assessed for eligibility by a study nurse. Eligible participant will then be taken through the consenting process. Participants whose parents have consented and have themselves assented when appropriate will then be randomized to either the influenza vaccine or placebo arm.

Schedule of follow up visits: After enrolment, each participant will be given a 6 month appointment for a review and a subsequent repeat of the TCDs. At the end of the 12 month follow up, each participant will at closure have repeat TCDs.

Blood investigations: At enrollment, blood will be drawn by venipuncture to assess for the inflammatory VCAM-1 and gene profile IL4R 503P locus, complete blood count panel, serum creatinine, serum urea and electrolytes, liver function tests.

Study visits: The study visits will include a baseline visit at enrollment, every 6 months and whenever the patient comes to the clinic or admitted at the pediatric emergence unit at Mulago National referral hospital. Patients who miss their scheduled study visits will be called within a week and actively followed to attend the visit before the month lapses. Patients who miss two consecutive study visits will be considered lost to follow up and attempts will be made to establish their current state as to whether they have a stroke.

Adverse effects monitoring: The participants will be counseled to report any untoward effect that they experience after receiving a study drug following GCP/ICH criteria. An adverse monitoring form will be completed for each study visit. Serious adverse effects that are potentially fatal or fatal will be reported to the ethics review board within 24hours of the occurrence of the adverse effect.

Local safety and data safety and monitoring committee: A data safety and monitoring committee will be set up to review the data so as to ascertain the continuous safety of the study drugs. This committee will comprise of a senior consultant pediatrician, biostatician and research scientist.

Stopping rules: There shall be no stopping rules Data Management: The principal investigator, co-investigator and clinical research nurses will have access to records.

Quality control and quality assurance: Data will be evaluated for compliance with protocol and accuracy in relation to source documents. The study will be conducted in accordance with procedures identified in the protocol. SOPs will be used at all clinical and laboratory sites.

Ethics/protection of human subjects: This protocol will be approved by Makerere University College of Health Sciences School of Medicine Research and Ethics Committee and the Uganda National Council of Science and Technology before this study commences. Consent shall be got from the parents and assent will be sought from the children above 8.

Informed Consent Process: Written informed consent will be obtained from the parents and assent sought from the children above 8 years of aged.. Parents will be provided with literature on the symptoms and signs of stroke in order to enable them return to the hospital.

Subject Confidentiality: All records will be kept in a locked filing cabinet, which is accessed only by the investigators and the study nurse(s). All computer entry and networking programs will be done with coded numbers and initials only. Only the investigators, the clinical monitor, the ethics committees or any other regulatory agencies, at the request of the collaborator will have access to the records. Every effort will be taken to maintain confidentiality.

The study protocol, documentation, data and all other information generated will be held in strict confidence. Clinical information will not be released without written permission of the parents, except as necessary for monitoring. No information concerning the study or the data will be released to any unauthorized third party, without prior written approval of the sponsor.

Data handling and record keeping The Principal Investigator will be the data manager with responsibility for receiving, entering, cleaning, querying, analysing and storing all data that accrues from the study. He will be responsible for linking the epidemiological and clinical data from the field and the clinic with the laboratory data from the immunology, haematology and genetics laboratories.

Study Records Retention: Essential documents will be retained until at least 2 years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or at least 2 years have elapsed since the formal discontinuation of clinical development of the investigational product. These documents will be retained for a longer period however if required by the applicable regulatory requirements or by an agreement with the sponsor. It is the responsibility of the sponsor to inform the investigator/institution as to when these documents no longer need to be retained

Protocol Deviations:The investigator will conduct the trial in compliance with the protocol agreed to by the sponsor and the regulatory authority and which was given approval by ethics. The investigator will sign the protocol to confirm agreement. In event of a deviation all relevant authorities will be informed.

Data analysis: Data will be entered using EPI info version 6.0.The primary end point will be the incidence of stroke at 12 month follow up. The incidence will be calculated as the number of new cases that have occurred during the given interval of time divided by the population at risk at the beginning of the time interval. Data will be analyzed using SPSS version 16 (SPSS Inc, Chicago, IL, USA). Both uni-variate analysis and bi-variate analysis will be done.

The primary analyses will be performed with an intention to treat with p <0.05 considered significant. . Survival analysis will be used to compare between the two groups. In order to assess for time to event, we shall construct Kaplan Meier survival curves. The outcomes will be compared using a log rank test to determine if differences are statistically significant. The relative risks will be calculated as the measures of association as well as absolute difference in the outcomes. Missing data will be recorded as missing and not analyse.

Conflict of interest: None

Collaborative agreements: None

Intended use of results:

Study findings will upon completion of the study be compiled into a report that will be copied or made available to the following: Nurture program, department of paediatrics and child health, Sir Albert cook library, the Sickle Cell Clinic, Ministry of Health. Findings will be presented in both local and international conferences. Manuscripts will also be prepared for publication in peer reviewed scientific journals.

Other information: The trial is not supported by another grant.

ELIGIBILITY:
Inclusion Criteria:

* • Age between 2 years and 12 years

  * All children whose parents will have consented and those above 7years will have to assent

Exclusion Criteria:

* • All children with previous strokes

  * Children who have acute illness and are not clinically stable
  * Any child with previous documented adverse event following immunization (AEFI).

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2018-08-22 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of stroke | 12 months
  • Incidence of stroke: The incidence of stroke is defined as the occurrence of a focal neurological deficit in a child lasting at least 24 hours if it has a vascular basis during the study period. Each child suspected to have stroke will have a brain cranial tomography (CT) scan done to confirm the diagnosis. This diagnosis will then be adjudicated by a team comprising of a pediatrician, neurologist and a radiologist.

SECONDARY OUTCOMES:
VCAM levels | 12
  • The levels of inflammatory markers VCAM-1 and gene profile IL4R 503P locus: blood will extracted from a participant by veni-puncture every 6 months and whenever a participant comes to the clinic when ill or is admitted.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of paediatrics and child Health,Makerere university, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No